CLINICAL TRIAL: NCT00280215
Title: Renal Protective Effect of ACEI and ARB in Primary Hyperoxaluria
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate number of patients, lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Dr. Dawn S. Milliner, Mayo Clinic, Rochester MN
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2203-05; NIH grant # DK 73354
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hyperoxaluria
Keywords: Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria; Hyperoxaluria, Primary | interventions — Angiotensin-Converting Enzyme Inhibitors; Lisinopril; Angiotensin Receptor Antagonists; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will be randomized to a combination of Angiotensin Converting Enzyme Inhibitor and Angiotensin Receptor Blocker. Patients will be randomized to a combination of ARB(losartan 50 mg daily in adult patients, 0.7 mg/kg/day in patients < 40 kg) ACE-I (lisinopril 10 mg daily in adult patients, 0.15 mg/kg/day in pediatric patients < 40 kg) to be taken for 24 months.
  Interventions: Drug: ACEI / Angiotensin converting enzyme inhibitor; Drug: ARB /Angiotensin Receptor Blocker
- 2 (Placebo Comparator): Patients will take placebo for 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACEI / Angiotensin converting enzyme inhibitor — Patients will be randomized to a combination of Angiotensin Converting Enzyme Inhibitor and Angiotensin Receptor Blocker, Patients will be randomized to a combination of ARB(losartan 50 mg daily in adult patients, 0.7 mg/kg/day in patients < 40 kg) ACE-I (lisinopril 10 mg daily in adult patients, 0.15 mg/kg/day in pediatric patients < 40 kg) to be taken for 24 months.
  Other Names: Lisinopril
  Arms: 1
Drug: ARB /Angiotensin Receptor Blocker — Patients will be randomized to a combination of Angiotensin Converting Enzyme Inhibitor and Angiotensin Receptor Blocker,Patients will be randomized to a combination of ARB(losartan 50 mg daily in adult patients, 0.7 mg/kg/day in patients < 40 kg) ACE-I (lisinopril 10 mg daily in adult patients, 0.15 mg/kg/day in pediatric patients < 40 kg) to be taken for 24 months.
  Other Names: Losartan
  Arms: 1
Drug: Placebo — Patients will receive placebo for 24 months
  Arms: 2

SUMMARY:
This study will test the effectiveness of two medications: ACEI (angiotensin converting enzyme inhibitor)and ARB (angiotensin receptor blocker) in reducing the renal injury induced by hyperoxaluria in patients with Primary Hyperoxaluria.

Hypothesis: Calcium oxalate crystal deposition in the kidney causes inflammation and resulting injury to kidney tissue. Angiotensin blockade will improve these changes, thus slowing the progression of renal insufficiency in patients with Primary Hyperoxaluria.

DETAILED DESCRIPTION:
In patients with primary hyperoxaluria (PH), deficiency of hepatic enzymes important in disposition of glyoxylate results in marked hyperoxaluria. Calcium oxalate crystals and high oxalate concentrations in the renal filtrate result in inflammation and injury in the renal parenchyma. Loss of renal function over time is characteristic, with end stage renal failure occurring in half the patients by age 35 years, but as early as infancy in some patients. Experience in animal models of hyperoxaluria, and from other renal diseases, supports a role for ACEI and ARB medications in ameliorating inflammation and injury thus providing a renal protective effect.

We propose to study the short-term effect of combined angiotensin converting enzyme inhibitor (ACEI) and angiotensin receptor blocking (ARB) therapy in patients with PH, in a controlled, randomized, two-year study. Primary endpoints will be urinary markers of renal tubular injury (retinol binding protein (RBP), alpha 1 microglobulin (α1m), γ-glutamyl transferase (GGT)) and interstitial fibrosis (transforming growth factor beta 1 (TGFβ1). Secondary endpoints will be the rates of change in renal tubular injury and renal function as determined by serum creatinine and creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PH established by liver enzyme analysis in the patient or an affected sibling, DNA testing for mutations of the AGXT and GR/HPR gene, or meeting clinical criteria (Urine oxalate > 70 mg/1.73 m2/day in the absence of malabsorption or dietary excess of oxalate. Elevated urine glycolate or glycerate provides supporting evidence of type I or type II PH, respectively).
2. Hyperoxaluria that persists during treatment with pyridoxine.
3. Ten years of age or older.
4. Glomerular filtration rate > 50 ml/min/1.73 m2 at the start of the study.
5. Women of child bearing age will be required to use adequate contraception for 3 months before and throughout the study.
6. Patients will be on a stable program of pyridoxine, neutral phosphate, or citrate medications -

Exclusion Criteria:

a. Age < 10 years. b. Glomerular filtration rate < 50 at start of study c. Hypersensitivity to ACEI or ARB medications d. Chronic use of ACEI or ARB medications prior to enrollment e. Hyperkalemia f. Previous renal transplant g. Homozygosity for the G170R mutation of AGXT h. Unwillingness to use adequate contraception during the study. i. Pregnancy

-

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Two-year change in the urinary markers of renal tubular injury and interstitial fibrosis | 2 years

SECONDARY OUTCOMES:
Rate of change in 1. Renal tubular injury markers and 2. Renal function as determined by serum creatinine and creatinine clearance. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dawn S Milliner, M.D., Principal Investigator — Mayo Clinic Hyperoxaluria Center, Rochester MN

REFERENCES:
- [Background] Milliner DS, Eickholt JT, Bergstralh EJ, Wilson DM, Smith LH. Results of long-term treatment with orthophosphate and pyridoxine in patients with primary hyperoxaluria. N Engl J Med. 1994 Dec 8;331(23):1553-8. doi: 10.1056/NEJM199412083312304. PMID 7969325
- [Background] Khan SR, Shevock PN, Hackett RL. Urinary enzymes and calcium oxalate urolithiasis. J Urol. 1989 Sep;142(3):846-9. doi: 10.1016/s0022-5347(17)38928-0. PMID 2570167
- [Background] Lieske JC, Monico CG, Holmes WS, Bergstralh EJ, Slezak JM, Rohlinger AL, Olson JB, Milliner DS. International registry for primary hyperoxaluria. Am J Nephrol. 2005 May-Jun;25(3):290-6. doi: 10.1159/000086360. Epub 2005 Jun 15. PMID 15961949
- [Background] Huang C, Kim Y, Caramori ML, Fish AJ, Rich SS, Miller ME, Russell GB, Mauer M. Cellular basis of diabetic nephropathy: II. The transforming growth factor-beta system and diabetic nephropathy lesions in type 1 diabetes. Diabetes. 2002 Dec;51(12):3577-81. doi: 10.2337/diabetes.51.12.3577. PMID 12453917
- [Background] Goumenos DS, Tsakas S, El Nahas AM, Alexandri S, Oldroyd S, Kalliakmani P, Vlachojannis JG. Transforming growth factor-beta(1) in the kidney and urine of patients with glomerular disease and proteinuria. Nephrol Dial Transplant. 2002 Dec;17(12):2145-52. doi: 10.1093/ndt/17.12.2145. PMID 12454225
- [Background] Scaglione R, Argano C, Parrinello G, Colomba D, Di Chiara T, Ferrante A, Di Garbo V, Avellone G, Licata G. Relationship between transforming growth factor beta1 and progression of hypertensive renal disease. J Hum Hypertens. 2002 Sep;16(9):641-5. doi: 10.1038/sj.jhh.1001465. PMID 12214261
- [Background] Abbate M, Zoja C, Rottoli D, Corna D, Tomasoni S, Remuzzi G. Proximal tubular cells promote fibrogenesis by TGF-beta1-mediated induction of peritubular myofibroblasts. Kidney Int. 2002 Jun;61(6):2066-77. doi: 10.1046/j.1523-1755.2002.00380.x. PMID 12028447
- [Background] Toblli JE, Ferder L, Stella I, Angerosa M, Inserra F. Protective role of enalapril for chronic tubulointerstitial lesions of hyperoxaluria. J Urol. 2001 Jul;166(1):275-80. PMID 11435885
- [Background] Toblli JE, Stella I, Angerosa M, Nyberg C, Ferder L, Inserra F: Transforming growth factor-b1 (TGF--b1) and collagen typ III in hyperoxaluric rats treated with enalapril. J Am Soc Nephrol 8:528A, 1997.
- [Background] Toblli JE, Stella I, de Cavanagh E, Angerosa M, Inserra F, Ferder L. Enalapril prevents tubulointerstitial lesions by hyperoxaluria. Hypertension. 1999 Jan;33(1 Pt 2):225-31. doi: 10.1161/01.hyp.33.1.225. PMID 9931109
- [Background] Danielpour D. Improved sandwich enzyme-linked immunosorbent assays for transforming growth factor beta 1. J Immunol Methods. 1993 Jan 14;158(1):17-25. doi: 10.1016/0022-1759(93)90254-5. PMID 8429213
- [Background] Sato M, Muragaki Y, Saika S, Roberts AB, Ooshima A. Targeted disruption of TGF-beta1/Smad3 signaling protects against renal tubulointerstitial fibrosis induced by unilateral ureteral obstruction. J Clin Invest. 2003 Nov;112(10):1486-94. doi: 10.1172/JCI19270. PMID 14617750
- [Background] Border WA, Noble NA. Interactions of transforming growth factor-beta and angiotensin II in renal fibrosis. Hypertension. 1998 Jan;31(1 Pt 2):181-8. doi: 10.1161/01.hyp.31.1.181. PMID 9453300
- [Background] Haugen EN, Croatt AJ, Nath KA. Angiotensin II induces renal oxidant stress in vivo and heme oxygenase-1 in vivo and in vitro. Kidney Int. 2000 Jul;58(1):144-52. doi: 10.1046/j.1523-1755.2000.00150.x. PMID 10886559
- [Background] de Cavanagh EM, Fraga CG, Ferder L, Inserra F. Enalapril and captopril enhance antioxidant defenses in mouse tissues. Am J Physiol. 1997 Feb;272(2 Pt 2):R514-8. doi: 10.1152/ajpregu.1997.272.2.R514. PMID 9124472
- [Background] Taal MW, Brenner BM. Renoprotective benefits of RAS inhibition: from ACEI to angiotensin II antagonists. Kidney Int. 2000 May;57(5):1803-17. doi: 10.1046/j.1523-1755.2000.00031.x. PMID 10792600
- [Background] Basile DP. The transforming growth factor beta system in kidney disease and repair: recent progress and future directions. Curr Opin Nephrol Hypertens. 1999 Jan;8(1):21-30. doi: 10.1097/00041552-199901000-00005. PMID 9914857
- [Background] Taal MW, Brenner BM. Combination ACEI and ARB therapy: additional benefit in renoprotection? Curr Opin Nephrol Hypertens. 2002 Jul;11(4):377-81. doi: 10.1097/00041552-200207000-00001. PMID 12105385
- [Background] Noda M, Matsuo T, Fukuda R, Ohta M, Nagano H, Shibouta Y, Naka T, Nishikawa K, Imura Y. Effect of candesartan cilexetil (TCV-116) in rats with chronic renal failure. Kidney Int. 1999 Sep;56(3):898-909. doi: 10.1046/j.1523-1755.1999.00614.x. PMID 10469358
- [Background] Akerstrom B, Logdberg L, Berggard T, Osmark P, Lindqvist A. alpha(1)-Microglobulin: a yellow-brown lipocalin. Biochim Biophys Acta. 2000 Oct 18;1482(1-2):172-84. doi: 10.1016/s0167-4838(00)00157-6. PMID 11058759
- [Background] Yu H, Yanagisawa Y, Forbes MA, Cooper EH, Crockson RA, MacLennan IC. Alpha-1-microglobulin: an indicator protein for renal tubular function. J Clin Pathol. 1983 Mar;36(3):253-9. doi: 10.1136/jcp.36.3.253. PMID 6186698
- [Background] Kirsztajn GM, Nishida SK, Silva MS, Ajzen H, Moura LA, Pereira AB. Urinary retinol-binding protein as a prognostic marker in glomerulopathies. Nephron. 2002 Apr;90(4):424-31. doi: 10.1159/000054730. PMID 11961401
- [Background] Norden AG, Scheinman SJ, Deschodt-Lanckman MM, Lapsley M, Nortier JL, Thakker RV, Unwin RJ, Wrong O. Tubular proteinuria defined by a study of Dent's (CLCN5 mutation) and other tubular diseases. Kidney Int. 2000 Jan;57(1):240-9. doi: 10.1046/j.1523-1755.2000.00847.x. PMID 10620205
- [Background] Westhuyzen J, Endre ZH, Reece G, Reith DM, Saltissi D, Morgan TJ. Measurement of tubular enzymuria facilitates early detection of acute renal impairment in the intensive care unit. Nephrol Dial Transplant. 2003 Mar;18(3):543-51. doi: 10.1093/ndt/18.3.543. PMID 12584277
- [Background] Werness PG, Brown CM, Smith LH, Finlayson B. EQUIL2: a BASIC computer program for the calculation of urinary saturation. J Urol. 1985 Dec;134(6):1242-4. doi: 10.1016/s0022-5347(17)47703-2. PMID 3840540
- [Background] Kavanagh JP, Jones L, Rao PN. Calcium oxalate crystallization kinetics studied by oxalate-induced turbidity in fresh human urine and artificial urine. Clin Sci (Lond). 2000 Feb;98(2):151-8. PMID 10657269
- [Background] Fan J, Chandhoke PS. Examination of crystalluria in freshly voided urines of recurrent calcium stone formers and normal individuals using a new filter technique. J Urol. 1999 May;161(5):1685-8. PMID 10210440
- [Background] Werness PG, Bergert JH, Smith LH: Crystalluria. J Crystal Growth 53:166-181, 1981
- See also: Mayo Clinic Hyperoxaluria Center home page — http://www.mayoclinic.org/nephrology-rst/hyperoxaluriacenter.html
- See also: The Oxalosis and Hyperoxaluria Foundation — http://www.ohf.org
- See also: Mayo Clinic Hyperoxaluria Center-disease information page — http://www.mayoclinic.org/hyperoxaluria/